CLINICAL TRIAL: NCT00443950
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of Etanercept in Chinese Subjects With Active Rheumatoid Arthritis Receiving Methotrexate
Brief Title: Study Evaluating the Efficacy and Safety of Etanercept in Chinese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A1-319
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis; Chinese
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The objective of this study is to compare in Chinese subjects with rheumatoid arthritis (RA) the efficacy and safety in this subject population of 50 mg once-weekly injections of etanercept versus placebo in subjects receiving methotrexate. This is a multi-center, double-blind, randomized, parallel and placebo-controlled outpatient study. Approximately 150 subjects will participate in this study for about 18 weeks including a screening period up to 4 weeks, 12-week treatment period, and a 2-week follow-up period at approximately 25 sites.

ELIGIBILITY:
Inclusion Criteria:

* Must be of Chinese ancestry and living in China.
* Meets the American Rheumatism Association 1987 Revised Criteria for the Classification of RA.
* Have active RA at the time of study enrollment (before the start of the screening period,) as demonstrated by 5 swollen and 5 tender/painful joints.

Exclusion Criteria:

* Previous receipt of etanercept; antibody to tumor necrosis factor (TNF) antibody (infliximab, adalimumab), anti-CD4 antibody or diphtheria IL-2 fusion protein (DAB IL-2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is ACR20 response at 12 weeks.

SECONDARY OUTCOMES:
Physician global assessments
Morning stiffness in minutes
Pain visual analog scale(VAS)
Health assessment questionnaire(HAQ)
C-reactive protein (CRP) values, Subject global assessments
Number of tender and swollen joints
ACR20 (at visit other than week 12)
ACR50
ACR70 responses

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (4):
- China (4):
  - Beijing
  - Guangzhou
  - Shanghai
  - Xi'an